CLINICAL TRIAL: NCT01331694
Title: Outcomes and Costs Associated With Initiating Maintenance Treatment With Fluticasone Propionate 250mcg/Salmeterol Xinafoate 50mcg Combination (FSC) Versus Anticholinergics Including Tiotropium (TIO) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112646
Record Dates: First submitted 2011-03-10; First posted 2011-04-08 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination; Tiotropium Bromide; Ipratropium; Albuterol; Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD: copd patients 65 years and older
  Interventions: Drug: fluticasone/salmeterol combination (FSC) 250/50mcg; Drug: tiotropium; Drug: ipratropium bromide alone or in fixed dose combination with albuterol

INTERVENTIONS:
Drug: fluticasone/salmeterol combination (FSC) 250/50mcg — patients initiating treatment with fluticasone/salmeterol combination (FSC) 250/50mcg
  Other Names: Advair (TM)
Drug: tiotropium — patients initiating treatment with tiotropium
  Other Names: Spiriva (TM)
Drug: ipratropium bromide alone or in fixed dose combination with albuterol — patients initiating treatment with ipratropium/albuterol
  Other Names: Atrovent (TM); Combivent (TM)

SUMMARY:
To evaluate COPD-related clinical outcomes and total healthcare utilization in commercially insured (at least 40 years with a subanalysis of those aged 65 years and older) COPD population associated with the use of fluticasone/salmeterol combination (FSC) 250/50mcg compared to other initial maintenance therapies (IMTs), specifically, tiotropium bromide (TIO), and either ipratropium bromide or ipratropium bromide/albuterol (IP).

This is a hypothesis testing study

Ho: There is no difference in time to first COPD-related events between FSC and TIO and FSC and IP Ha: There is a difference in time to first COPD-related events between FSC and TIO and FSC and IP

Hypothesis for the key secondary outcome of COPD-related costs that was tested was:

Ho: There is no difference in COPD-related costs between FSC and TIO and FSC and IP Ha: There is a difference in COPD-related costs between FSC and TIO and FSC and IP

DETAILED DESCRIPTION:
All population i.e. at least 40 years: Each initial maintenance treatment (IMT) cohort (FSC 250/50mcg dose only, IP, and TIO) includes patients aged 40 years and older with at least 9 months of continuous enrollment (6 months pre-index and at least three months post-index) with a primary or secondary diagnosis of COPD [International Classification of Disease, 9th revision, Clinical Modification (ICD-9-CM) codes 491.xx, 492.xx or 496.xx]. Patients are observed such that everyone provides minimum 6 months of pre index baseline data and minimum 3 months post index (risk analysis) and minimum 12 months post index for cost analysis. Patients must receive either a 30-day supply of FSC or IP or TIO as the initial IMT medication, indicating "intent to treat." Patients may not also have a prescription filled for the other IMT medication within 60 days of the index date, or for the combination therapy budesonide/ formoterol (BFC), an inhaled corticosteroid (ICS) or a long acting beta agonist (LABA). Six months of observation (continuous enrollment) prior to the index date is assessed to confirm that the patient meets the inclusion and exclusion criteria as well as to identify baseline characteristics and covariates. Cost analysis was done using a 12 months fixed follow up period. Outcome measures are assessed during the post-index period

Elderly cohort 65+: Identical methods and design were used for subanalyses in patients aged 65 years and over except comparison was FSC vs. TIO only.

75+ cohort: Identical methods and design were used for subanalyses in patients aged 75 years and over except comparison was FSC vs. TIO only.

ELIGIBILITY:
Inclusion Criteria -

IMT Cohorts (subjects selected by order of criteria)

* claim for one of the study medications and must not receive another study medication within 60 days of the initial maintenance therapy, indicating "intent to treat."
* at least one COPD-related ED or one COPD-related hospitalization, or two COPD-related outpatient visits (OV) associated with primary or secondary diagnosis for COPD (ICD-9-CM code 491.xx, 492.xx or 496.xx), at any time during the observation period (July 1, 2005 through June 30, 2008) in the database.
* Aged 65+ years on the index date or aged 40 and over for the sub-analysis.
* Continuous enrollment in a health plan for at least 6 months prior (pre-index) to initiation of IMT and at least three months after the first initiation of IMT (post-index).
* at least one prescription claim in the pre-index and each year of the post-index period for which they have follow-up.

Exclusion Criteria - All Cohorts

* primary or secondary diagnosis of respiratory tract cancer (larynx, trachea, or pleura). (ICD-9-CM codes 161, 161.X, 162, 163, 163.X, 231, 231.X).
* In the pre-index period, no claims for any of the cohort IMT medications, nor for any other Advair or budesonide/formoterol fixed dose combination, FSC combination medications, and may only have respiratory medication pharmacy claims for drugs included in the pre-index severity of illness assessment (Methylxanthines, Leukotriene Modifiers/Inhibitors, Omalizumab and Mast Cell Stabilizers).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All population i.e. U>U40 years: Each initial maintenance treatment (IMT) cohort (FSC 250/50mcg dose only, IP, and TIO) includes patients aged 40 years and older with at least 9 months of continuous enrollment (6 months pre-index and at least three months post-index) with a primary or secondary diagnosis of COPD [International Classification of Disease, 9th revision, Clinical Modification (ICD-9-CM) codes 491.xx, 492.xx or 496.xx]. Patients are observed such that everyone provides minimum 6 months of pre index baseline data and minimum 3 months post index (risk analysis) and minimum 12 months post index for cost analysis. Patients must receive either a 30-day supply of FSC or IP or TIO as the initial IMT medication, indicating "intent to treat." Patients may not also have a prescription filled for the other IMT medication within 60 days of the index date, or for the combination therapy budesonide/ formoterol (BFC), an inhaled corticosteroid (ICS) or a long acting beta agonist (LABA).
Sampling Method: Non-Probability Sample
Enrollment: 76130 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Dalal AA, Roberts MH, Petersen HV, Blanchette CM, Mapel DW. Comparative cost-effectiveness of a fluticasone-propionate/salmeterol combination versus anticholinergics as initial maintenance therapy for chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2010 Dec 31;6:13-22. doi: 10.2147/COPD.S15455. PMID 21311689

RESULTS

PARTICIPANT FLOW:
Groups:
- Risk Population: FSC: Participants in the Overall Risk Population (participants with 3-12 months of follow-up after initial treatment arm prescription) receiving fluticasone propionate/salmeterol combination (FSC) 250 micrograms (mcg)/50 mcg
- Risk Population: IP: Participants in the Overall Risk Population (participants with 3-12 months of follow-up after initial treatment arm prescription) receiving ipratropium bromide 18 mcg or ipratropium bromide/albuterol 18 mcg/103 mcg (IP)
- Risk Population: TIO: Participants in the Overall Risk Population (participants with 3-12 months of follow-up after initial treatment arm prescription) receiving tiotropium bromide (TIO) 18 mcg
- Cost Population: FSC: Participants in the Overall Cost Population (participants with 12 months of follow-up after initial treatment arm prescription) receiving fluticasone propionate/salmeterol combination (FSC) 250 mcg/50 mcg
- Cost Population: IP: Participants in the Overall Cost Population (participants with 12 months of follow-up after initial treatment arm prescription) receiving ipratropium bromide 18 mcg or ipratropium bromide/albuterol 18 mcg/103 mcg (IP)
- Cost Population: TIO: Participants in the Overall Cost Population (participants with 12 months of follow-up after initial treatment arm prescription) receiving tiotropium bromide (TIO) 18 mcg
Period: Overall Study
Arm/Group | Risk Population: FSC | Risk Population: IP | Risk Population: TIO | Cost Population: FSC | Cost Population: IP | Cost Population: TIO
Started | 16684 | 14449 | 12659 | 12595 | 10617 | 9126
Completed | 16684 | 14449 | 12659 | 12595 | 10617 | 9126
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risk Population: FSC: Participants in the Overall Risk Population (participants with 3-12 months of follow-up after initial treatment arm prescription) receiving fluticasone propionate/salmeterol combination (FSC) 250 mcg/50 mcg
- Total: Total of all reporting groups
Arm/Group | Risk Population: FSC | Risk Population: IP | Risk Population: TIO | Cost Population: FSC | Cost Population: IP | Cost Population: TIO | Total
Number analyzed (Participants) | 16684 | 14449 | 12659 | 12595 | 10617 | 9126 | 76130
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at initial treatment arm prescription
  Years | 62.8 (12.00) | 65.2 (12.59) | 64.5 (11.33) | 62.8 (11.92) | 65.0 (12.42) | 64.5 (11.34) | 64.0 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender reported in claims records
  Participants
    Female | 9127 | 7143 | 5862 | 6914 | 5298 | 4256 | 38600
    Male | 7557 | 7306 | 6797 | 5681 | 5319 | 4870 | 37530

OUTCOME MEASURES:

1. Primary Outcome: Time to First Chronic Obstructive Pulmonary Disease (COPD) Event
Description: The first COPD event occurring after 30 days from initial treatment arm prescription was measured. Four categories of COPD events were analyzed; either a hospitalization or emergency department visit; an emergency department visit; an outpatient visit followed by an oral corticosteroid prescription claim within 10 days; an outpatient visit followed by an oral antibiotic prescription claim within 10 days.
Time Frame: Anytime from 30 days to 12 months after initial treatment arm prescription
Population: All participants from a large database comprised of information from enrollment files and facility, professional service, and outpatient pharmacy claims from a variety of private healthcare benefit plans covering over 40 million patients enrolled in over 70 health plans (providing data continuously) across the United States.
Measure: Mean (Standard Error); unit: days
Groups:
- Risk Population TIO: Participants in the Overall Risk Population (participants with 3-12 months of follow-up after initial treatment arm prescription) receiving tiotropium bromide (TIO) 18 mcg
Arm/Group | Risk Population: FSC | Risk Population: IP | Risk Population TIO
Number analyzed (Participants) | 16684 | 14449 | 12659
days
  Hospitalization or emergency department visit | 325.17 (0.39) | 315.89 (0.56) | 321.59 (0.51)
  Emergency department visit | 330.24 (0.28) | 324.47 (0.43) | 328.48 (0.37)
  Outpatient visit with oral steroid fill | 332.74 (0.22) | 328.23 (0.31) | 331.23 (0.30)
  Outpatient visit with antibiotic fill | 329.96 (0.30) | 326.73 (0.39) | 326.70 (0.39)
Statistical Analysis 1: Comparison: Risk Population: FSC vs Risk Population: IP; Test type: Superiority or Other; Hazard Ratio (HR) = 1.64, 95% CI [1.50 to 1.79] — Hazard ratio for hospitalization or emergency department visit for IP compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization
Statistical Analysis 2: Comparison: Risk Population: FSC vs Risk Population TIO; Test type: Superiority or Other; Hazard Ratio (HR) = 1.29, 95% CI [1.17 to 1.41] — Hazard ratio for hospitalization or emergency department visit for TIO compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization
Statistical Analysis 3: Comparison: Risk Population: FSC vs Risk Population: IP; Test type: Superiority or Other; Hazard Ratio (HR) = 1.78, 95% CI [1.59 to 2.00] — Hazard ratio for emergency department visit for IP compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization
Statistical Analysis 4: Comparison: Risk Population: FSC vs Risk Population TIO; Test type: Superiority or Other; Hazard Ratio (HR) = 1.33, 95% CI [1.17 to 1.51] — Hazard ratio for emergency department visit for TIO compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization
Statistical Analysis 5: Comparison: Risk Population: FSC vs Risk Population: IP; Test type: Superiority or Other; Hazard Ratio (HR) = 1.65, 95% CI [1.41 to 1.94] — Hazard ratio for outpatient visit with oral steroid fill for IP compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization
Statistical Analysis 6: Comparison: Risk Population: FSC vs Risk Population TIO; Test type: Superiority or Other; Hazard Ratio (HR) = 1.49, 95% CI [1.26 to 1.76] — Hazard ratio for outpatient visit with oral steroid fill for TIO compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization
Statistical Analysis 7: Comparison: Risk Population: FSC vs Risk Population: IP; Test type: Superiority or Other; Hazard Ratio (HR) = 1.39, 95% CI [1.23 to 1.57] — Hazard ratio for outpatient visit with antibiotic fill for IP compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization
Statistical Analysis 8: Comparison: Risk Population: FSC vs Risk Population TIO; Test type: Superiority or Other; Hazard Ratio (HR) = 1.33, 95% CI [1.17 to 1.51] — Hazard ratio for outpatient visit with antibiotic fill for TIO compared to FSC; HR estimate adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization

2. Secondary Outcome: Average Annual Adjusted Post-Index COPD-Related Costs
Description: Medical costs are associated with COPD-related medical care (claims submitted with a primary International Classification of Diseases, 9th Revision, Clinical Modification diagnosis of COPD) and pharmaceutical care (treatment arm medications, oral corticosteroids, oral antibiotics, short-acting beta-agonists, long-acting beta-agonists [LABA], inhaled corticosteroids [ICS], ICS/LABA combinations, etc.. Means are adjusted for age, sex, geographic region, pre-initial treatment comorbidities, and COPD-related utilization. Total costs are the sum of medical care and pharmacy costs.
Time Frame: Incurred over the 12 month period after initial treatment arm prescription
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Cost Population: FSC | Cost Population: IP | Cost Population: TIO
Number analyzed (Participants) | 12595 | 10617 | 9126
United States dollars
  Medical | 1076 (1119) | 2481 (2770) | 1419 (1572)
  Pharmacy | 972 (175) | 614 (225) | 985 (355)
  Total | 2068 (1190) | 2841 (1858) | 2408 (1511)

ADVERSE EVENTS:
Description: This study was a retrospective observational study; thus, no serious adverse events or adverse events were collected.
Arm/Group | Risk Population: FSC | Risk Population: IP | Risk Population: TIO | Cost Population: FSC | Cost Population: IP | Cost Population: TIO
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.